CLINICAL TRIAL: NCT01728597
Title: Optimization of Non-contrast Enhanced 1.5 Tesla and 3 Tesla Cardiac Magnetic Resonance Imaging Techniques and Acquisition of Normal Values
Brief Title: Non-contrast Enhanced Cardiac Magnetic Resonance Normal Values and Imaging Protocols
Acronym: CMR-TECH
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Amt der Steiermärkischen Landesregierung, Abteilung 3 (Unknown)
Responsible Party: Principal Investigator, Ursula Reiter, PhD, Medical University of Graz
Other Study IDs: CMR-12-TECH-02
Record Dates: First submitted 2012-11-03; First posted 2012-11-20 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: no history of cardiovascular diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- healthy volunteers: MR compliant volunteers with no history of cardiovascular diseases

SUMMARY:
One of the main problems in cardiac magnetic resonance (MR) investigations is the strong dependence of the achieved image quality on optimal settings of sequence parameters and anatomical and physiological situations and it is well known that the diagnostic impact of cardiac MR investigations crucially depends on the adaption of imaging protocols to patients' state and ability to cooperate.

The aim of the present study is the evaluation and optimization of various 1.5 Tesla and 3 Tesla cardiac MR investigation protocols without application of contrast agent as well as the acquisition of normal values for new cardiac MR images techniques:

* normal myocardial morphology: T1-, T2- and T2*-weighted imaging and acquisition of normal values of magnetic relaxation times (sequence- and protocol dependent),
* normal cardiac function: systolic and diastolic function (sequence- and protocol dependent),
* cardiac anatomy and coronary artery imaging: feasibility to evaluate length, diameter and blood flow (sequence- and protocol dependent),
* normal blood flow topologies in the heart and the surrounding great vessels: 2D- and 3D blood flow imaging and evaluation techniques (sequence- and protocol dependent).

ELIGIBILITY:
Inclusion Criteria:

* No history of cardiac or pulmonary diseases
* ability to give informed consent

Exclusion Criteria:

* General MR exclusion criteria eg. patients with metal devices or other magnetic material in or on the subjects body which will be hazardous for MR investigation (e.g. heart pace-maker, brain aneurysm clip, nerve stimulators, electrodes, penile implants, coloured contact lenses, patch to deliver medications through the skin, any metal implants as rods, joints, plates, pins, screws, nails or clips, embolization coil, or any metal fragments or shrapnel in the body),
* pregnancy,
* claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
cardiac volumes | up to 1 week
  volumes of cardiac chambers in the cardiac cycle [ml], sequence- and protocol dependent
cardiac performance | up to 1 week
  ejection fraction of cardiac chambers [%], sequence- and protocol dependent
cardiac muscle mass | up to 1 week
  systolic and end-diastolic mass of cardiac chambers [g], sequence- and protocol dependent
coronary artery anatomy | up to 1 week
  length and diameter [mm], sequence-, and protocol dependent
blood flow velocity | up to 1 week
  maximum, minimum and average velocity [cm/s], sequence-, and protocol dependent
blood flow vorticity | up to 1 week
  number of vortices of blood flow in the heart and surrounding great vessels, sequence and protocol dependent
blood flow timing | up to 1 week
  time points of characteristic blood flow patterns in the heart and surrounding great vessels in the cardiac cycle [ms], sequence-, and protocol dependent
magnetic relaxation times | up to 1 week
  systolic and diastolic T1, T2, T2* [ms], sequence- and protocol dependent

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Reiter, PhD, Principal Investigator — Medical Unitersity Graz, Department of Radiology, Division of General Radiology
Locations (1):
- Medical Unitersity Graz, Department of Radiology, Division of General Radiology, Graz, Styria, Austria

REFERENCES:
- [Result] Reiter U, Reiter G, Dorr K, Greiser A, Maderthaner R, Fuchsjager M. Normal diastolic and systolic myocardial T1 values at 1.5-T MR imaging: correlations and blood normalization. Radiology. 2014 May;271(2):365-72. doi: 10.1148/radiol.13131225. Epub 2013 Dec 6. PMID 24475837
- [Result] Krauter C, Reiter U, Reiter C, Nizhnikava V, Masana M, Schmidt A, Fuchsjager M, Stollberger R, Reiter G. Automated mitral valve vortex ring extraction from 4D-flow MRI. Magn Reson Med. 2020 Dec;84(6):3396-3408. doi: 10.1002/mrm.28361. Epub 2020 Jun 18. PMID 32557819
- [Result] Reiter C, Reiter U, Krauter C, Nizhnikava V, Greiser A, Scherr D, Schmidt A, Fuchsjager M, Reiter G. Differences in left ventricular and left atrial function assessed during breath-holding and breathing. Eur J Radiol. 2021 Aug;141:109756. doi: 10.1016/j.ejrad.2021.109756. Epub 2021 May 7. PMID 34023727
- [Result] Reiter C, Reiter G, Krauter C, Scherr D, Schmidt A, Fuchsjager M, Reiter U. Evaluation of left ventricular and left atrial volumetric function from native MR multislice 4D flow magnitude data. Eur Radiol. 2024 Feb;34(2):981-993. doi: 10.1007/s00330-023-10017-3. Epub 2023 Aug 15. PMID 37580598
- [Result] Gillette K, Gsell MAF, Prassl AJ, Karabelas E, Reiter U, Reiter G, Grandits T, Payer C, Stern D, Urschler M, Bayer JD, Augustin CM, Neic A, Pock T, Vigmond EJ, Plank G. A Framework for the generation of digital twins of cardiac electrophysiology from clinical 12-leads ECGs. Med Image Anal. 2021 Jul;71:102080. doi: 10.1016/j.media.2021.102080. Epub 2021 Apr 22. PMID 33975097